CLINICAL TRIAL: NCT06664541
Title: Decision-Making and Quality of Life Surrounding Hematologic Disease and Gene Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00007772
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Transfusion Dependent Beta Thalassemia; Sickle Cell Disease
Keywords: quality of life
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients or parents of pediatric patients diagnosed with beta-thalassemia or sickle cell disease and eligible to receive treatment for their disease with gene therapy.

SUMMARY:
Determine knowledge, attitudes, and beliefs among adult patients, and parents of pediatric patients, with transfusion dependent beta-thalassemia and sickle cell disease toward gene therapy to treat their or their child's illness, and to assess the likely impact of gene therapy on patients' quality of life.

DETAILED DESCRIPTION:
The overarching aim of this research is to determine knowledge, attitudes, and beliefs among adult patients, and parents of pediatric patients, with transfusion dependent beta-thalassemia toward gene therapy to treat their or their child's disease, and to assess the likely impact of gene therapy on patients' quality of life. We will compare and contrast these findings to those obtained from a sample of adult patients and parents of pediatric patients with sickle cell disease. We will also assess perceptions of the pros/cons of gene therapy, including its financial and time costs.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (ages 18+) or parents of pediatric patients (<age 18) eligible to receive treatment for their disease with gene therapy

Exclusion Criteria:

* Non-English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (ages 18+) or parents of pediatric patients (<age 18) diagnosed with transfusion-dependent beta thalassemia or sickle cell disease and eligible to receive treatment for their disease with gene therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Past 12 months
  Health related quality of life is measured by a modified patient reported outcome measure, the Transfusion-dependent Quality of Life (TranQoL) assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States